CLINICAL TRIAL: NCT05454826
Title: Investigation of the Effect of Cold Application in Addition to Relaxation Exercises in Patients with Migraine
Brief Title: Investigation of the Effect of Cold Application in Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eylül Pınar KISA (Other)
Responsible Party: Sponsor-Investigator, Eylül Pınar KISA, Dr., Biruni University
Organization: Biruni University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: migraine
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Migraine; Cold; Relaxation; Exercise
MeSH Terms: conditions — Migraine Disorders; Common Cold; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cold application group (Experimental): applied relaxation exercise+ cold pack
  Interventions: Other: Cold Application
- control group (Experimental): applied relaxation exercise
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — 1st group (n=15) relaxation exercises, 2nd group (n=15) relaxation exercises+cold compression. The exercise program will be applied for 6 weeks, 3 days a week * 45 minutes. Relaxation exercises will be applied to the patients 3 days a week using web-based methods (Zoom).
  Other Names: Relaxation exercise applications
  Arms: control group
Other: Cold Application — 1st group (n=15) relaxation exercises, 2nd group (n=15) relaxation exercises+cold compression. The exercise program will be applied for 6 weeks, 3 days a week * 45 minutes. Relaxation exercises will be applied to the patients 3 days a week using web-based methods (Zoom).
  Other Names: Relaxation exercise+ cold pack applications
  Arms: Cold application group

SUMMARY:
Migraine is a headache that is paroxysmal and can last for hours, sometimes even days due to untreated or ineffective treatment is usually unilateral, throbbing, severe enough to prevent the person's daily life activities, and increases with head movements. It is a chronic disorder characterized by recurrent moderate and severe headaches, mostly associated with a few symptoms in the autonomic nervous system. Migraine consists of recurrent headache attacks accompanied by neurological, gastrointestinal, and autonomic symptoms.

Migraine is the most common chronic headache in epidemiological studies. Studies have shown that migraine affects 12% of the general population. The aim of migraine treatment is to reduce the frequency, duration, and severity of migraine attacks, to reduce the losses caused by migraine, and increase the quality of life.

In the treatment of migraine, non-pharmacological treatment is as important as pharmacological treatment. Some individuals prefer drug-free treatment methods because of the side effects drugs. In recent years, as the mechanisms of headaches have been better understood, significant developments have been made in treatment methods. Different physiotherapy and rehabilitation methods have been used for treatment. There are studies in which cold application is used in migraine patients, but a study evaluating the effectiveness of cold application has not been found in the literature. The systemic effects of cold have two main purposes: to maintain the current body temperature and to produce energy to raise the fallen body temperature. Knowing both the local and systemic effects of cold guides its use in treatment. The aim of this study was to diagnose migraine.

To investigate the effectiveness of cold application applied in addition to relaxation exercises in individuals.

DETAILED DESCRIPTION:
Thirty migraine patients diagnosed by a physician will be included in our study.

Participants will be divided into two groups as randomized controlled. Only relaxation exercises will be applied to a group for 6 weeks, 3 days a week. In the other group, relaxation In addition to the exercises, cold will be applied. The sociodemographic information of the patients will be evaluated with the "patient case form", the pain severity will be evaluated with the "visual analog scale" and the quality of life will be evaluated with the world health organization quality of life scale ('whoqol-bref').

Migraine disability rating scale (MIDAS) will be used for functionality. Statistical analysis of data SPSS It will be done using the 24.0 (Statistical Package for Social Sciences) program and p≤0.05 will be considered statistically significant in all analyzes.

The reason why the investigators chose cold application in addition to relaxation exercises in our study is that it is a low-cost, risk-free method that everyone can access. It is also an easy-to-apply method.

ELIGIBILITY:
Inclusion Criteria:

* be between 20-45 years old
* Having been diagnosed with migraine at least 6 months ago
* Patient's ability to use a computer

Exclusion Criteria:

* Being in the period of menstruation
* Sensitivity to cold (those who have 5 or more sensitivity on a 10 cm scale)
* Having any neurological or orthopedical problems
* Using antidepressants etc.
* Poor mental state

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Migraine Disability Assessment questionnaire | 0-6. week
  The Migraine Disability Assessment questionnaire (MIDAS) questionnaire was developed to measure the effect of headaches on a person's daily functioning. MIDAS takes into account the last three months and consists of five questions. It is a simple and short survey. These questions are used to determine your score and are then matched to a disability level. As the score increases, the severity of migraine pain increases.

SECONDARY OUTCOMES:
World Health Organization quality of life scale ('whoqol-bref') | 0-6. week
  The scale measures physical, mental, social and environmental well-being and consists of 26 questions. The scale was used in patients with migraine. Since each domain independently expresses the quality of life in its own field, field scores are calculated between 4-20.
  The higher the score, the higher the quality of life.
Visual Analog Scale | 0-6. week
  Patients will be asked to mark the degree of pain they feel during the attack period and during the attack-free period on the 10 cm VAS line. "If you wanted to rate your headache, how many points would you give it? 10 if you have very severe pain; If you have no pain, mark 0 points." The marked point will be measured and recorded with a tape measure.
Patient case form | 0-6. week
  It consists of questions of age, gender, height, weight and body mass index, educational status, alcohol/cigarette use, history of other diseases, family history of migraine, history of accident and trauma, medications used, number of attacks in the last 1 month, and duration of attacks. . In this form, the person's sensitivity to cold will also be questioned.

CONTACTS AND LOCATIONS:
Locations (1):
- Eylül Pınar Kısa, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided